CLINICAL TRIAL: NCT00314470
Title: Image and Dosimetry Related Research of Department of Medical Physics, Cross Cancer Institute
Status: Completed | Type: Observational
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: EX-0001/ethics 21312
Record Dates: First submitted 2006-04-11; First posted 2006-04-14 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2012-04

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to retrospectively have access to image files of patients.

ELIGIBILITY:
Inclusion Criteria:

* Subject 18 years of age and over

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Representative selection from the database (images) of clinical research patients approved for other protocols.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2006-01; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gino Fallone, PhD, Principal Investigator — AHS Cancer Control Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada